CLINICAL TRIAL: NCT02360150
Title: Evaluation of Myocardial Viability in Late Presentation Myocardial Infarction: Dual Energy Cardiac CT vs. Cardiac MRI.
Brief Title: Evaluation of Myocardial Viability : Dual Energy Cardiac CT vs. Cardiac MRI
Acronym: InfarctusGSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2013/205/HP
Record Dates: First submitted 2014-12-15; First posted 2015-02-10 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Myocardial Infarction
Keywords: cardiac angiography; cardiac MRI
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- second propeller arm scanner (Experimental): The experimental procedure is to conduct a second helical scanner strictly centered on the heart, 10 minutes after the first helix without inject contrast medium, to assess late enhancement to the inclusion visit.
  Interventions: Radiation: second propeller arm scanner

INTERVENTIONS:
Radiation: second propeller arm scanner — The experimental procedure is to conduct a second helical scanner strictly centered on the heart, 10 minutes after the first helix without inject contrast medium, to assess late enhancement.

SUMMARY:
The purpose of this study is therefore to show that associated with cardiac angiography echocardiography, in myocardial seen late, would provide the information necessary for the decision revascularization, in a timely manner.

This would allow the patient to avoid duplication of tests including risk related to coronary angiography (bleeding complications, stroke ...) and those related to the implantation of coronary stent (stent) without expected earnings in case of non-viability . This would also reduce the length of hospital stay and costs due to numerous reviews.

DETAILED DESCRIPTION:
Percutaneous coronary intervention is not recommended in stable patients with late presentation myocardial infarction, and myocardial viability needs to be evaluated before the procedure. The aim of the study is to evaluate the sensibility and specificity of dual-energy CT for the evaluation of myocardial viability in comparison to cardiac MRI.

The experimental procedure is limited to a second CT acquisition performed 10 minutes in dual energy mode.

Sensitivity and Specificity of delayed enhancement >50% of myocardial thickness provided by dual-energy CT will be evaluated in comparison to cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Major patient
* Patient with electrical, biological and clinical signs of myocardial infarction, with late presentation (>24 hours)
* Creatinine clearance (calculated using the Cockcroft (<age 65) or MDRD (> 65 years))formula > 30 ml / min.
* Affiliation to the french social security scheme.
* Women of childbearing age: Negative pregnancy test (urine test).
* Postmenopausal women, menopause confirmation of diagnosis
* Patient able to understand the spoken and written French.
* Signature of informed consent

Exclusion Criteria:

* Collapsus or organ failure requiring urgent care in intensive care unit
* Arrhythmia and/or non-reducible tachycardia.
* History of allergic reaction after iodinated contrast medium injection.
* History of nephrogenic systemic fibrosis.
* History of claustrophobia
* Unbalanced asthma.
* Acute pulmonary edema.
* Pregnant or breastfeeding women.
* Clinical signs of thyrotoxicosis.
* Person placed under judicial protection,
* Patient suffering from serious psychiatric disease.
* Patients participating in another clinical trial.
* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Number of patient with a possible evaluation of myocardial viability using dual-energy cardiac CT | Day 4
  To study the sensitivity of dual-energy cardiac CT for the evaluation of myocardial viability, in patients with late presentation myocardial infarction.

SECONDARY OUTCOMES:
Number of patient with a possible evaluation of myocardial viability using cardiac MRI | Day 4
  To study the sensitivity of cardiac MRI for the evaluation of myocardial viability in patients with late presentation myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin DUBOURG, Doctor, Principal Investigator — University Hospital, Rouen; Jean-Nicolas DACHER, Professor, Study Director — University Hospital, Rouen
Locations (1):
- University Hospital of Rouen, Rouen, Normandy, France